CLINICAL TRIAL: NCT03150615
Title: Effect of Enteral Nutrition on Delayed Gastric Emptying After Pancreaticoduodenectomy: A Prospective, Randomized Controlled Trial
Brief Title: Enteral Nutrition After Pancreaticoduodenectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Yi Miao, Prof., Director of Pancreas Center, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NMU-JSPH-PC-Nutrition
Record Dates: First submitted 2017-03-26; First posted 2017-05-12 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Cancer of Pancreas; Cancer of Duodenum; Ampulla of Vater Cancer; Cholangiocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms; Duodenal Neoplasms; Cholangiocarcinoma | interventions — Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Early enteral nutrition (Experimental): Nasojejunal tube insertion was done intraopratively. Early enteral nutrition with standard enteral formulas administered through the nasojejunal tube. Oral intake was encouraged as long as the patient can tolerate.
  Interventions: Other: Early enteral nutrition; Device: nasojejunal tube insertion; Other: Oral intake
- Saline Group (Placebo Comparator): Nasojejunal tube insertion was done intraopratively. Saline was administered through the nasojejunal tube. Oral intake was encouraged as long as the patient can tolerate.
  Interventions: Other: Saline; Device: nasojejunal tube insertion
- ERAS Group (Other): Nasojejunal tube insertion was done intraopratively. None was administered through the nasojejunal tube. Oral intake was encouraged as long as the patient can tolerate.
  Interventions: Device: nasojejunal tube insertion; Other: Oral intake

INTERVENTIONS:
Other: Early enteral nutrition — Naso-jejunal tube will be placed intraoperatively. The distal end of the feeding tube would be placed at 30 cm distal to Treitz ligament. Standard enteral diet, administered through a nasojejunal tube, is started on the 1st postoperative day and increased daily by 20-40 ml up to the estimated level.
  After PD, enteral nutrition liquid regimen will be used step by step from postoperative day 1 to postoperative day 7.Patients are targeted to receive calories for 25 kcal/kg/day. Meanwhile, oral food intake was not restricted.
  Arms: Early enteral nutrition
Other: Saline — Naso-jejunal tube will be placed intraoperatively. The distal end of the feeding tube would be placed at 30 cm distal to Treitz ligament.
  After PPPD,Only Normal Saline were given through nasojejunal tube. Entral nutrition was not administrated. Patients intake food orally at will.
  Arms: Saline Group
Device: nasojejunal tube insertion
  Other Names: Naso-jejunal tube will be placed intraoperatively.
Other: Oral intake — Patients was encouraged to drink water on postoperative day 1, to eat liquid diet on postoperative day 2, to eat semi-solid on postoperative day 3, to eat solid food on postoperative day 4.
  Arms: ERAS Group; Early enteral nutrition

SUMMARY:
Pancreaticoduodenectomy (PD) is the treatment of choice for resectable periampullary cancer. PD is still associated with a relatively a high incidence of delayed gastric emptying. And, there are no acknowledged strategies to avoid DGE. Several feeding strategies have been investigated to cope with this problem. However, there is still no consensus concerning the best nutrition support method after pancreaticoduodenectomy. The purpose of this study is to determine the effect of nutrition support methods on DGE after pancreaticoduodenectomy: early enteral nutrition or total parenteral nutrition.

Patients undergoing pancreatoduodenectomy will be randomized to receive early enteral nutrition (EN group), or Saline administration (Saline group), or oral intake only (Natural control). The EN group will receive standard enteral diet administered through a nasojejunal tube. Enteral nutrition will be started on the 1st postoperative day and increased daily by 20-40 ml up to the estimated level. The Saline group will receive saline administered through a nasojejunal tube beginning from the 1st postoperative day. Oral intake will not be restricted in all three group.

ELIGIBILITY:
Inclusion Criteria:

Patients underwent selective pancreaticoduodenectomy Patients ≥18 years old and ≤80 years old Having given written informed consent

Exclusion Criteria:

Previous gastric resection or intestinal reconstruction Preoperative complete parenteral or enteral feeding ASA score ≥4 Pregnant women Severe malnutrition Patient who cannot give written informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-09; Primary Completion 2017-12 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Incident rate of delayed gastric emptying | 30 days
  DGE represents the inability to return to a standard diet by the end of the first postoperative week and includes prolonged nasogastric intubation of the patient. Three different grades (A,B,and C) were defined based on the impact on the clinical course and on postoperative management by ISGPS.

SECONDARY OUTCOMES:
Postoperative hospital stay length | 60 days
Overall morbidity rate | 30 days
Postoperative mortality rate | 30 days
Rehospitalization rate | 60 days
Infectious complications | 30 days
Evaluation of the severity of the complications | 30 days
  according to classification of Dindo-Clavien
Pancreatic fistulas | 30 days
  evaluation of the occurrence of pancreatic fistulas, grade B and C, in both groups of patients
Hemorrhagic complications | 30 days
  evaluation of the occurrence of hemorrhagic complications, grade B and C, in both groups of patients
Maximum Plasma Concentration fasting plasma GLP-1 level | Preoperative day 1, Postoperative day 1, Postoperative day 4, Postoperative day 7
  Fasting plasma concentration GLP-1 level was monitored

CONTACTS AND LOCATIONS:
Overall Officials: Yi Miao, Prof., Principal Investigator — Pancreas Center, The First Affiliated Hospital of Nanjing Medical University; Junli Wu, MD,PhD, Study Director — Pancreas Center, The First Affiliated Hospital of Nanjing Medical University; Jishu Wei, MD,PhD, Principal Investigator — Pancreas Center, The First Affiliated Hospital of Nanjing Medical University
Locations (1):
- The first affiliated hospital of Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Shen Y, Jin W. Early enteral nutrition after pancreatoduodenectomy: a meta-analysis of randomized controlled trials. Langenbecks Arch Surg. 2013 Aug;398(6):817-23. doi: 10.1007/s00423-013-1089-y. Epub 2013 May 22. PMID 23695769
- [Background] Lu JW, Liu C, Du ZQ, Liu XM, Lv Y, Zhang XF. Early enteral nutrition vs parenteral nutrition following pancreaticoduodenectomy: Experience from a single center. World J Gastroenterol. 2016 Apr 14;22(14):3821-8. doi: 10.3748/wjg.v22.i14.3821. PMID 27076767
- [Background] Zhu XH, Wu YF, Qiu YD, Jiang CP, Ding YT. Effect of early enteral combined with parenteral nutrition in patients undergoing pancreaticoduodenectomy. World J Gastroenterol. 2013 Sep 21;19(35):5889-96. doi: 10.3748/wjg.v19.i35.5889. PMID 24124335
- [Background] Perinel J, Mariette C, Dousset B, Sielezneff I, Gainant A, Mabrut JY, Bin-Dorel S, Bechwaty ME, Delaunay D, Bernard L, Sauvanet A, Pocard M, Buc E, Adham M. Early Enteral Versus Total Parenteral Nutrition in Patients Undergoing Pancreaticoduodenectomy: A Randomized Multicenter Controlled Trial (Nutri-DPC). Ann Surg. 2016 Nov;264(5):731-737. doi: 10.1097/SLA.0000000000001896. PMID 27429039
- [Background] Rayar M, Sulpice L, Meunier B, Boudjema K. Enteral nutrition reduces delayed gastric emptying after standard pancreaticoduodenectomy with child reconstruction. J Gastrointest Surg. 2012 May;16(5):1004-11. doi: 10.1007/s11605-012-1821-x. Epub 2012 Jan 19. PMID 22258876
- [Derived] Liu X, Chen Q, Fu Y, Lu Z, Chen J, Guo F, Li Q, Wu J, Gao W, Jiang K, Dai C, Miao Y, Wei J. Early Nasojejunal Nutrition Versus Early Oral Feeding in Patients After Pancreaticoduodenectomy: A Randomized Controlled Trial. Front Oncol. 2021 Apr 29;11:656332. doi: 10.3389/fonc.2021.656332. eCollection 2021. PMID 33996579